CLINICAL TRIAL: NCT01959113
Title: Phase 1 Study of the Short-term Antimicrobial Action of Transplanted Bacteria in Adult Patients With Atopic Dermatitis
Brief Title: Validation of the Short-term Antimicrobial Action of Transplanted Bacteria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Richard Gallo, Professor and Chair, Division of Dermatology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSD 131244.1
Record Dates: First submitted 2013-09-30; First posted 2013-10-09 (Estimated); Results first posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Atopic Dermatitis
Keywords: Microbiome; Bacteria transplant; Atopic dermatitis treatments
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous Microbiome Transplant (Experimental): Each individual's autologous microbiome transplant cream will be applied to one of their arms. This arm is the treatment arm.
  Interventions: Biological: Autologous Microbiome Transplant
- Placebo Arm (Placebo Comparator): This arm will have a base moisturizer alone applied to it during the third visit.
  Interventions: Other: Placebo Arm

INTERVENTIONS:
Biological: Autologous Microbiome Transplant
  Arms: Autologous Microbiome Transplant
Other: Placebo Arm
  Other Names: The placebo arm will have a commercially available moisturizer applied to it.
  Arms: Placebo Arm

SUMMARY:
Unlike healthy control skin, the skin of patients with atopic dermatitis (AD) is frequently colonized by Staphylococcus aureus (S. aureus), putting these patients at increased risk of S. aureus skin infections. In addition, research in the investigator's lab has shown that these patients have fewer protective antimicrobial Staphylococcal species such as Staphylococcal epidermidis (S. epidermidis) that are known to produce antimicrobial peptides that play a role in protecting the skin from invading pathogens. In this study, the investigator will attempt to decrease S. aureus colonization and increase colonization by protective Staph species in AD patients. First the investigator will capture the bacteria on subjects' lesional AD skin. Next the investigator will selectively grow the subject's antimicrobial Staphylococcal colonies and place them into a base moisturizer. The moisturizer plus bacteria will be applied to one of the subject's arms, and the moisturizer alone (without bacteria) to the other arm. The investigator will then do a quantitative wash of the bacteria growing on each arm one day later in order to determine whether the S. aureus abundance was affected by the application of the transplanted bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are not pregnant or lactating
* 18-80 years of age
* Diagnosis of atopic dermatitis for at least 6 months using the Hanifin and Rajka Diagnostic Criteria for atopic dermatitis
* Presence of lesional atopic dermatitis skin in both antecubital fossae
* Positive methicillin-sensitive S. aureus colonization based on results of a skin culture taken from one of their AD-affected antecubital fossae during the screening visit

Exclusion Criteria:

* Use of any topical AD treatments (including topical steroids, topical calcineurin inhibitors) to either arm within one week of either screening visit
* Use of any oral/systemic AD therapies (antihistamines, steroids) within 28 days of either screening visit
* Severe AD that would worsen significantly from holding a participant's usual topical/oral AD medications for the time periods required in the inclusion/exclusion criteria (one week prior to the screening visits and during the study for topical medications and 28 days prior to screening visits and during the study for oral medications)
* Subjects who have taken a bleach bath within a week prior to screening, or who take bleach baths during the study
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Subjects with Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier
* Any subject who is immunocompromised (e.g. provides researchers with a history lymphoma, HIV/AIDS, Wiskott-Aldrich Syndrome) or has a history of malignant disease (with the exception of non-melanomatous skin cancer). This information will be gathered verbally from the patient while taking a medical history from the patient, and will not involve further testing such as an HIV test.
* Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
* Active bacterial, viral or fungal skin infections
* Any noticeable breaks or cracks in the skin on either arm, including severely excoriated skin or skin with open or weeping wounds suggestive of an active infection or increased susceptibility to infection.
* Ongoing participation in another investigational trial
* Use of any oral or topical antibiotic for up to four weeks prior to screening
* Use of any systemic immunosuppressive therapy (e.g. cyclosporin, methotrexate, etc.) within four weeks of screening.
* Sensitivity to or difficulty tolerating Dove fragrance-free bar soap, Dial antibacterial liquid soap, Cetaphil lotion, or alcohol-based cleaners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Division of Dermatology, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with AD were recruited from the University of California, San Diego (UCSD), La Jolla, CA, and the National Jewish Health (NJH), Denver, CO.
Pre-assignment Details: All subjects avoided any treatments and therapies that may potentially affect skin microbiome before sample collection.
Units Other Than Participants: arms
Groups:
- Autologous Microbiome Transplant and Placebo (Split-design): Each individual's autologous microbiome transplant cream will be applied to one of their arms. This arm is the treatment arm.
  Autologous Microbiome Transplant
  Placebo vehicle cream will be applied to the contralateral arm. This arm is the placebo arm.
Period: Overall Study
Arm/Group | Autologous Microbiome Transplant and Placebo (Split-design)
Started | 5; 10 arms
Completed | 5; 10 arms
Not Completed | 0; 0 arms

BASELINE CHARACTERISTICS:
Population: 5 subjects with AD were enrolled in the study. Each of the subject's arms was randomly assigned to treatment with AMT or placebo.
Arm/Group | Autologous Microbiome Transplant and Placebo (Split-design)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (2.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Relative Staphylococcus Aureus Abundance
Description: The technique of quantitative washes will be used to determine the Staphylococcus aureus abundance on an area of lesional AD skin on the subject's forearm as a ratio of baseline S. aureus abundance
Time Frame: 24-hours post-transplant
Measure: Mean (Standard Deviation); unit: ratio to baseline S. aureus abundance
Units Other Than Participants: arms
Groups:
- Placebo Arm: This arm will have a base moisturizer alone applied to it during the third visit.
  Placebo Arm
- Autologous Microbiome Transplant: Each individual's autologous microbiome transplant cream will be applied to one of their arms. This arm is the treatment arm.
  Autologous Microbiome Transplant
Arm/Group | Placebo Arm | Autologous Microbiome Transplant
Number analyzed (Participants) | 5 | 5
Number analyzed (arms) | 5 | 5
ratio to baseline S. aureus abundance | 0.13 (0.2) | 12.2 (10.1)

ADVERSE EVENTS:
Time Frame: 30 days after baseline visit
Description: Participants were asked about adverse events by phone 30 days after baseline visit.
Groups:
- Placebo (Split-design): Placebo vehicle cream will be applied to the contralateral arm. This arm is the placebo arm.
Arm/Group | Autologous Microbiome Transplant | Placebo (Split-design)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Microbiome Transplant (N=5) | Placebo (Split-design) (N=5)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes